CLINICAL TRIAL: NCT02406716
Title: Semaphorins 3A and 4D Levels in Heart Failure Patients: Pathogenesis and Clinical Correlation
Brief Title: Semaphorins 3A and 4D Levels in Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: NW-2401-ZV
Record Dates: First submitted 2015-03-29; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HF: Heart failure patients
  Interventions: Other: Biospecimen retention
- Controls: Healthy donors
  Interventions: Other: Biospecimen retention

INTERVENTIONS:
Other: Biospecimen retention

SUMMARY:
This study hypothesis is that Semaphorins 3A and 4D levels are overexpressed in patients with heart failure. Study protocol:

Hospitallized patients with new onset or previously diagnosed heart failure will be recruited to the study. Control group will include healthy people with no medical records or chronic treatment at the same age range. After signing an informed constent form, full medical history and blood samples will be collected. A second blood sample will be collected 8 weeks later, assuming the patient was discharged and not hospitalized since than. The blood samples will be analyzed by Bnai Zion Medical Center Immunology labs for the above semaphorins levels in the heart failure group and control group. Statistical analysis will then commence for possible correlatoion with different clinical parameters.

DETAILED DESCRIPTION:
In few previous published studies, Semaphorins 3A levels are overexpressed in patients with heart failure. The aim of our study is the compare semaphorin 3A and 4D in patients with acute decompansated heart failure with healthy donors. Second aim is to compare semaphorin level in the same patients in time of hospitalization and few weeks later when the heart failure presumingly controled. Statistical analysis will then commense for possible correlatoion with different clinical parameters like NYHA (new york heart association) status of the patient, lenghts of hospitalization and BNP (brain natriuretic peptide) levels at time of admition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new onset or previously diagnosed heart failure.
* Heart failure diagnosis can be based on clinical judgment, echocardiography or elevated BNP levels

Exclusion Criteria:

* Patients with acute myocardial infarction diagnosed clinicly and labratory

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with new onset or previously diagnosed heart failure
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Semaphrone 3A and 4D levels | one year

SECONDARY OUTCOMES:
BNP level | one year
  Brain natriuretic peptide level in patient plasma

CONTACTS AND LOCATIONS:
Overall Officials: Zahava Vadas, MD. PHD., Principal Investigator — Bnai Zion Medical Center, Immunology devision